CLINICAL TRIAL: NCT07362667
Title: A Prospective, Multicenter, Observational Cohort Study on the Efficacy and Safety of Bronchoscopic Airway Clearance and Amphotericin B Spraying in Patients With Allergic Bronchopulmonary Aspergillosis
Brief Title: A Study of the Efficacy and Safety of Bronchoscopic Airway Clearance and Amphotericin B Spraying in Patients With ABPA
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Prof., Qianfoshan Hospital
Other Study IDs: ABPA-001
Record Dates: First submitted 2025-12-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: ABPA; Allergic Bronchopulmonary Aspergillosis; Allergic Bronchopulmonary Aspergillosis (ABPA); Airway Clearance; Mucus Plug; Amphotericin B; Bronchoscope
Keywords: Allergic Bronchopulmonary Aspergillosis; ABPA; Amphotericin B; bronchoscope; Airway Clearance; mucus plug
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, sputum, bronchoalveolar lavage fluid, urine, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: The observation group was treated with standard drug therapy (oral glucocorticoids combined or not combined with oral antifungal drugs), combined with bronchoscopic airway clearance and amphotericin B spraying treatment
  Interventions: Procedure: The patients were treated with bronchoscopic airway clearance and amphotericin B spraying
- Control group: Control group: The control group was treated with standard drug therapy (oral glucocorticoids with or without oral antifungal drugs). The previous treatment for bronchial asthma was maintained, including inhaled corticosteroids + long-acting β-receptor agonists, leukotriene receptor antagonists, etc.

INTERVENTIONS:
Procedure: The patients were treated with bronchoscopic airway clearance and amphotericin B spraying — In addition to standard medical therapy (oral glucocorticoids with or without oral antifungal agents), bronchoscopic airway clearance and bronchoscopic spraying of amphotericin B (depending on the effectiveness of bronchoscopic mucus plug removal, At least one time of bronchoscopic airway clearance and amphotericin B spraying). The previous treatment for bronchial asthma was maintained, including inhaled corticosteroids + long-acting β-receptor agonists, leukotriene receptor antagonists, etc.
  Groups: Observation group

SUMMARY:
To evaluate the efficacy and safety of bronchoscopic airway clearance and amphotericin B spraying in the treatment of allergic bronchopulmonary aspergillosis

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of allergic bronchopulmonary aspergillosis, according to the ISHAM guidelines for the diagnosis and treatment of allergic bronchopulmonary aspergillosis (2024 revision), and the presence of mucus plugs or hyperattenuated mucus confirmed by chest high-resolution CT (HRCT).
2. Active disease: Newly diagnosed allergic bronchopulmonary aspergillosis or an acute exacerbation after discontinuation of treatment (defined as a > 14 day history of clinical worsening or radiographic progression of allergic bronchopulmonary aspergillosis and a ≥50% increase in total serum IgE from the last recorded value during the stable phase, excluding other causes of the acute exacerbation) in patients with previously diagnosed allergic bronchopulmonary aspergillosis.
3. Age ≥ 18 years old.

Exclusion Criteria:

1. Allergic bronchopulmonary aspergillosis - serotype (i.e., meets the diagnostic criteria for allergic bronchopulmonary aspergillosis, but chest CT shows no obvious abnormality);
2. Patients with absolute or relative contraindications to electronic bronchoscopy;
3. Known history of allergy to amphotericin B or any of its excipients;
4. Patients with bronchiectasis caused by human immunodeficiency virus infection, active tuberculosis, pulmonary malignant tumor or other non-allergic bronchopulmonary aspergillosis;
5. Combined with other diseases requiring long-term systemic use of glucocorticoids or immunosuppressants (such as autoimmune diseases);
6. Patients with previous or current smoking history;
7. Pregnant or lactating women;
8. Currently participating in other interventional clinical research;
9. Any other conditions considered by the investigator to preclude participation in the study (e.g., nonadherence, predicted survival <1 year, or severe mental illness that prevented cooperation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with allergic bronchopulmonary aspergillosis included patients with newly diagnosed allergic bronchopulmonary aspergillosis and patients with acute exacerbation of allergic bronchopulmonary aspergillosis after drug withdrawal.
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic response rate after 4 months of treatment | 4 months
  Radiographic remission: defined as the removal of mucus plugs in the airway on radiographic examination
Immunological remission rate after 4 months of treatment | 4 months
  Immunological remission: defined as at least a 50% decrease in total serum IgE from baseline
The remission rate of clinical symptoms after 4 months of treatment | 4 months
  Clinical symptom relief: The semi-quantitative rating of clinical symptoms was evaluated using Likert scores with at least 50% improvement in symptoms

SECONDARY OUTCOMES:
Number of acute exacerbations within 1 year of drug withdrawal after 4 months of treatment | 1 year
Number of acute exacerbations within 2 years after 4 months of treatment | 2 years
Treatment response rate at 8 weeks | 8 weeks
Number of hospitalizations due to acute exacerbations of allergic bronchopulmonary aspergillosis | 2 years
Time from discontinuation to first exacerbation | 2 years
After drug withdrawal, the number of patients who achieved treatment remission | 2 years
  The remission phase was defined as sustained (>6 months) clinical-radiologic improvement in the absence of (or discontinuation of) glucocorticoid therapy and the absence of an increase in total serum IgE of 50% or more from the last recorded value during the stable phase
Quality of life score (AQLQ or mini-AQLQ) | 2 years
Serum total IgE | 2 years
All-cause mortality | 2 years
psychological Scale (Hospital Anxiety and Depression Scale, HADS) | 2 years
Aspergillus fumigatus sIgE | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No